CLINICAL TRIAL: NCT05909488
Title: Role of Umbilical Cord-derived Stem Cell Transplantation and Conditioned Medium to Inhibit Vision Loss in Retinitis Pigmentosa Phase I/II
Brief Title: Role of UC-MSC and CM to Inhibit Vision Loss in Retinitis Pigmentosa Phase I/II
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT/RP/06/2022
Record Dates: First submitted 2023-03-14; First posted 2023-06-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Allogeneic Mesenchymal Stem Cell; Umbilical Cord Mesenchymal Stem Cell; Conditioned Medium; Allogeneic Umbilical Cord Mesenchymal Stem Cell
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EYESTEM 001-X (Experimental): 1.8 ml cell preparations are suspended in Conditioned Media (CM) until it reaches a 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) suspension will be injected into the peribulbar.
  Interventions: Biological: 1.5 x 10^6 UC-MSC + CM
- EYESTEM 001-XF (Experimental): 1.8 ml cell preparations are suspended in Conditioned Media (CM) until it reaches a 2 ml volume of cell suspension. Umbilical Cord Mesenchymal Stem Cell (UC-MSC) suspension will be injected into the peribulbar.
  Interventions: Biological: 5 x 10^6 UC-MSC + CM

INTERVENTIONS:
Biological: 1.5 x 10^6 UC-MSC + CM — 1.5 million cells of UC-MSC in 2 ml of Conditioned Medium (CM)
  Arms: EYESTEM 001-X
Biological: 5 x 10^6 UC-MSC + CM — 5 million cells of UC-MSC in 2 ml of Conditioned Medium (CM)
  Arms: EYESTEM 001-XF

SUMMARY:
The study will perform UC-MSCs and CM transplantation. There are two groups with different dosages. The first group will be transplanted with 1.5 million cells, meanwhile, the second group is 5 million cells. Each group consists of 30 subjects. All groups will be transplanted via the peribulbar route. All groups will be observed until six months.

DETAILED DESCRIPTION:
The eyes we will give the transplant should be given an aseptic and antiseptic technique to prevent contamination from the inside and outside. Sterile cover attached to other parts of the face except for the eyes. 1.8 ml Umbilical Cord-derived Mesenchymal Stem Cell (UC-MSC) preparations are suspended in Conditioned Medium (CM) until it reaches a 2 ml volume of cell suspension. Two dosages will be prepared, 1.5 million and 5 million of UC-MSC. Stem cell suspension will be injected by peribulbar, and patients will be given a quinolone antibiotic if the injection is done. On day 1st and day 7th after therapy, patients will be observed the presence of infection, inflammation, and increased eye pressure. On day 7th, day 30th, and day 90th after therapy, patients will do a visual field test, visual acuity test, electroretinography, funduscopy, and Optical Coherence Tomography examination. The observations will be written in the table and analyzed by a statistic.

ELIGIBILITY:
Inclusion Criteria:

* Visus more than 20/100
* Have more than 0.68 uV on conical receptor cell amplitude checked by ERG
* Visual field equivalent diameter more than 10o
* Willing to sign informed consent as research subjects
* Willing to do the peribulbar injection with mesenchymal stem cells isolated from umbilical cord tissue
* Willing to do visual field checks with Humphrey's perimetry, vision tests with Snellen boards, Optical Coherent Tomography (OCT) examinations, electroretinogram examinations, and fill out a quality of life questionnaire

Exclusion Criteria:

* Pregnant or nursing women
* Positive result of HIV test
* Have a history of eye tumors
* Under immunosuppressive treatment or other drugs that can affect the growth of transplanted stem cells
* Have another eye disease such as diabetic retinopathy, uveitis, cataract, and glaucoma
* Do not come to control according to the schedule determined by the researcher (loss to follow up)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incident of Adverse Events | 1 day after injection
  assessment of infection, inflammation, eye pressure and patients complaints
Incident of Adverse Events | 1 week after injection
  assessment of infection, inflammation, eye pressure and patients complaints
Frequency of Adverse Events | 1 day after injection
  assessment of infection, inflammation, eye pressure and patients complaints
Frequency of Adverse Events | 1 week after injection
  assessment of infection, inflammation, eye pressure and patients complaints
Visual Acuity Test | 1 week after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Acuity Test | 1 month after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Acuity Test | 3 months after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Acuity Test | 6 months after injection
  a test to see the sharpness of vision using Snellen Chart which is read at a distance of 6 meters. Normal eye test results are stated in 6/6.
Visual Field Test | 1 week after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humphrey's perimetry.
Visual Field Test | 1 month after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humphrey's perimetry.
Visual Field Test | 3 months after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humphrey's perimetry.
Visual Field Test | 6 months after injection
  a test to assess the breadth of views of the lateral, medial, superior and inferior aspects using Humphrey's perimetry.
Funduscopy | 1 week after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Funduscopy | 1 month after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Funduscopy | 3 months after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Funduscopy | 6 months after injection
  an examination to see and assess the abnormalities and conditions in the ocular fundus using an ophthalmoscope. This examination is carried out by an ophthalmologist.
Electrorectinography | 1 week after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Electrorectinography | 1 month after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Electrorectinography | 3 months after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Electrorectinography | 6 months after injection
  an examination to provide a picture of objectivity, a quantitative measure of retinal function to monitor the function of stem cells and ganglion cells in the eye. This examination is carried out by a trained ophthalmologist.
Optical Coherence Tomography (OCT) | 1 week after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities.
Optical Coherence Tomography (OCT) | 1 month after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities.
Optical Coherence Tomography (OCT) | 3 months after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities.
Optical Coherence Tomography (OCT) | 6 months after injection
  is a diagnostic test that give the information about posterior segment structure, which is retina and optic nerve papillae so that it can be used to assess macular abnormalities.

SECONDARY OUTCOMES:
Patients Quality of Life | 1 week after injection
  Patient's quality of life using National Eye Institute-Visual Functional Questioner 25
Patients Quality of Life | 1 month after injection
  Patient's quality of life using National Eye Institute-Visual Functional Questioner 25
Patients Quality of Life | 3 months after injection
  Patient's quality of life using National Eye Institute-Visual Functional Questioner 25
Patients Quality of Life | 6 months after injection
  Patient's quality of life using National Eye Institute-Visual Functional Questioner 25
Pain evaluation | 6 months after injection
  Evaluation on level of pain felt by patients
Eye bump | 6 months after injection
  Evaluation on appearance of eye bump

CONTACTS AND LOCATIONS:
Overall Officials: dr. Muhammad B Sasongko, Sp.M, M.Epid, PhD, Principal Investigator — Gadjah Mada University, Faculty of Medicine; Cosmos Mangunsong, Doctor, Study Chair — Jakarta Eye Center; dr. Rifa Widyaningrum, M.Sc, PhD, Study Chair — Sardjito Hospital
Locations (1):
- RSUP Dr. Sardjito, Yogyakarta, DI Yogyakarta, Indonesia